CLINICAL TRIAL: NCT02288208
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose, Safety, Tolerability and Pharmacokinetics Study of Birinapant in Subjects With Chronic Hepatitis B
Brief Title: Phase I Safety and Tolerability Study of Birinapant in Chronic Hepatitis B
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to cranial nerve palsies observed
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TL32711-POC-0095-PTL
Record Dates: First submitted 2014-11-03; First posted 2014-11-11 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; entecavir; birinapant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antiviral Therapy & Birinapant (Experimental): Antiviral therapy (tenofovir 300 mg or entecavir 0.5 mg) taken once daily by mouth, and birinapant administered as a 30 minute IV infusion once weekly for four weeks.
  Interventions: Drug: Antiviral Therapy (tenofovir or entecavir); Drug: Birinapant
- Antiviral Therapy & Placebo (Placebo Comparator): Antiviral therapy (tenofovir 300 mg or entecavir 0.5 mg) taken once daily by mouth, and placebo (for birinapant) administered as a 30 minute infusion once weekly for four weeks.
  Interventions: Drug: Antiviral Therapy (tenofovir or entecavir); Drug: Placebo (for birinapant)

INTERVENTIONS:
Drug: Antiviral Therapy (tenofovir or entecavir)
Drug: Birinapant
  Arms: Antiviral Therapy & Birinapant
Drug: Placebo (for birinapant)
  Arms: Antiviral Therapy & Placebo

SUMMARY:
This study evaluates the addition of birinapant in subjects with chronic Hepatitis B who are currently receiving anti-viral therapy with either tenofovir or entecavir. Patients will receive either birinapant or placebo in addition to their anti-viral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of chronic Hepatitis B infection currently being treated with tenofovir or entecavir for at least 3 months
* Measurable titer of HBsAg
* HBV DNA level < 2 log copies/mL or 10² copies/mL
* No more than Child-Pugh score of 5 plus a valid FibroScan® of at least 10 readings with a median score of <7 and interquartile range of < 30%
* Adequate liver function, aspartate AST and ALT ≤2 x ULN
* Adequate renal function as evidenced by creatinine ≤2 mg/dL

Exclusion Criteria:

* Participation in any interventional study within 4 weeks prior to Screening
* Known HIV infection, Hepatitis C, or other significant hepatic disorder including cirrhosis (Child-Pugh Class B or C)
* Serious illness or autoimmune disease or other known liver disease
* Uncontrolled hypertension
* Impaired cardiac function, uncontrolled cardiac arrhythmias despite medications, or clinically significant cardiac disease
* Currently breast feeding, pregnant or planning on becoming pregnant
* Known allergy or hypersensitivity to any of the formulation components of birinapant or placebo, including citric acid
* History of cranial nerve palsy
* Current treatment with anti-TNF therapies or has received treatment with anti-TNF therapies within the last 6 months
* Use of non-steroidal anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From Screening through end of study, up to 13 weeks

SECONDARY OUTCOMES:
Pharmacokinetics of birinapant (in plasma): maximum concentration (Cmax), time of maximum concentration (Tmax), area under the curve (AUC) extrapolated to time infinity, AUC from dosing to last quantifiable concentration | Day -1 through Day 26
Pharmacokinetics of birinapant (in plasma): terminal elimination half-life (t1/2), clearance (CL), terminal disposition rate constant,volume of distribution (Vdss) | Day -1 through Day 26
Pharmacokinetics of oral antiviral medication (tenofovir or entecavir): Cmax, Tmax, AUC from dosing to last quantifiable concentration, t1/2, CL, terminal disposition rate constant, Vdss | Day -1, Day 1 and Day 22
Hepatitis B markers (Determine levels of HBsAg, HBeAg, HBV DNA, and HBsAb) | Screening through Day 29
  Determine levels of HBsAg, HBeAg, HBV DNA, and HBsAb
Pharmacodynamic effect of birinapant on cIAP1 and cIAP2 levels in peripheral blood mononuclear cells (PBMC) and levels of cluster of differentiation 4 and 8 (CD4+, CD+8) lymphocytes | Screening through Day 29

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - CMAX / Royal Adelaide Hospital, Adelaide, South Australia
  - Nucleus Network Limited / AMREP Precinct, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia